CLINICAL TRIAL: NCT00310362
Title: Use of Telehealth In-Home Messaging to Improve GI Endoscopy Completion Rates
Brief Title: Use of Telehealth In-home Messaging to Improve GI (Gastrointestinal) Endoscopy Completion Rates
Acronym: GIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 03-295
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
Keywords: telephone; telemedicine; mass screening; patient education; Patient compliance
MeSH Terms: conditions — Colorectal Neoplasms; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care with nurse phone call (Experimental): Usual Care--Nurses telephoned patients 7 days prior to appointment to remind patients about scheduled GI appointment and to answer any questions.
  Interventions: Behavioral: Use of Interactive Voice Response (IVR) system to improve adherence to GI appointments and prep procedures
- interactive voice response 3 days prior (Experimental): Interactive voice response system was used to remind patients 3 days before a scheduled appointment and to educate them about preparation procedures for the appointment (IVR3)
  Interventions: Behavioral: Use of Interactive Voice Response (IVR) system to improve adherence to GI appointments and prep procedures
- interactive voice response 7 days prior (Experimental): Interactive voice response system was used to remind patients 7 days before a scheduled appointment and to educate them about preparation procedures for the appointment (IVR7)
  Interventions: Behavioral: Use of Interactive Voice Response (IVR) system to improve adherence to GI appointments and prep procedures

INTERVENTIONS:
Behavioral: Use of Interactive Voice Response (IVR) system to improve adherence to GI appointments and prep procedures — Interactive voice response system (IVR) calls patients 7 or 3 days prior to their appointment. Information available in the IVR system is based on the same template nurses use in usual care and includes an appointment reminder, preparation instructions, basic information about the procedure, and answers to commonly asked questions.

SUMMARY:
Low endoscopy completion rates are a major problem in the VA, causing delay or failure to receive essential care, increased clinic wait times, lost capacity, increased costs, thus limiting endoscopic screening for colorectal cancer. This study tests whether an Interactive Voice Response (IVR) messaging system is equally effective in promoting the completion of flexible sigmoidoscopy and colonoscopy as usual clinical care practices that include phone calls from nurses to patients prior to preparation and procedures. Previous studies have examined the role of scheduling facilitation or patient adherence on endoscopy completion and the use of IVR technology to enhance patient adherence in other medical contexts. This is the first study, however, to evaluate the use of IVR for endoscopy completion and the first to compare it to the effectiveness of phone calls from nurses prior to an endoscopy appointment.

DETAILED DESCRIPTION:
Background:

Low endoscopy completion rates are a major problem nationwide and in the VA. For clinics, delays or failure to complete exams can cause clinic inefficiencies, such as increased wait times for needed procedures, lost capacity, and increased costs. For patients, delays reduce the chance for recommended timely screening consistent with practice guidelines and for diagnostic tests, can cause significant anxiety, delayed treatment and possibly poorer prognosis. This study tests whether an Interactive Voice Response (IVR) messaging system is equally effective in motivating patients to complete a flexible sigmoidoscopy or colonoscopy as usual clinical care practices, which include reminder phone calls from clinic nurses. This is the first study to evaluate the use of IVR for endoscopy completion and the first to compare it to the effectiveness of phone calls from nurses prior to an endoscopy appointment.

Objectives:

The primary set of objectives was to test whether IVR messaging was equivalent to clinic usual care (UC) practices in motivating patients to attend a scheduled flexible sigmoidoscopy or colonoscopy appointment and to adequately prepare for the exam. Secondary objectives included comparing patient satisfaction with UC and IVR phone calls and assessing if IVR or UC was more effective for sub-groups that may have more difficulty with preparation, including those with poor physical and mental functioning, health literacy, social support and trust in physicians and those with spinal cord injury, paraplegia, PTSD, or with little intention to be tested for colorectal cancer in the future.

Methods:

This was a stratified 3-arm randomized controlled trial among patients with upcoming flexible sigmoidoscopy or colonoscopy appointments. All patients who had a colonoscopy or flexible sigmoidoscopy appointment scheduled from August 20, 2007 through October 31, 2008 were assessed for inclusion in this study. Patients were not considered eligible if, based on a medical record review prior to randomization, they had unreliable means of receiving the intervention or the intervention would have provided inappropriate or inaccurate information. The three study arms included: 1) UC (nurse phone call 7 days prior to the procedure); 2) IVR7 (call from IVR system 7 days prior to procedure); and, 3) IVR3 (call from IVR system 3 days prior to procedure). One week after the initial appointment self-administered surveys were sent to all participants to assess satisfaction with reminder/motivation calls. Appointment and gastrointestinal (GI) procedure data were extracted from medical record files to assess study outcomes. The principal outcome measures were (1) attendance at the scheduled endoscopy appointment; (2) adequate preparation for the exam; (3) patient satisfaction with reminder/motivation telephone calls.

Status:

Complete

ELIGIBILITY:
Inclusion Criteria:

All patients with either flexible sigmoidoscopy or colonoscopy appointments scheduled greater than 7 days before their appointment in the GI endoscopy clinic from August 20, 2007 through October 31, 2008.

Exclusion Criteria:

Patients were not considered eligible for inclusion in the study if, based on a medical record review prior to randomization, they had unreliable means of receiving the intervention or the intervention would have provided inappropriate or inaccurate information. These patients included those who lived in a nursing or group home or homeless shelter; had no listed telephone number; scheduled the appointment less than 8 days in advance; or, had Type 1 diabetes, dementia or Alzheimer's or multiple GI procedures on the same day (such as those with both upper and lower GI procedures). All patients excluded from the study were assigned to usual care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3610 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan M. Griffin, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Griffin JM, Hulbert EM, Vernon SW, Nelson D, Hagel EM, Nugent S, Baines Simon A, Bangerter A, van Ryn M. Improving endoscopy completion: effectiveness of an interactive voice response system. Am J Manag Care. 2011 Mar;17(3):199-208. PMID 21504256

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care included nurse phone calls to participants 7 days prior to the scheduled appointment. Calls were intended as appointment reminders and opportunities for education on preparation procedures.
- IVR3: Arm 2 (IVR3) included interactive voice response calls delivered to patients 3 days prior to the scheduled appointment. Calls were intended as appointment reminders and as interactive, but pre-recorded, opportunities for education on preparation procedures.
- IVR7: Arm 3 (IVR7) included interactive voice response calls delivered to patients 7 days prior to the scheduled appointment. Calls were intended as appointment reminders and as interactive, but pre-recorded, opportunities for education on preparation procedures.
Period: Overall Study
Arm/Group | Usual Care | IVR3 | IVR7
Started | 1199 | 1205 | 1206
Completed | 1199 | 1205 | 1206
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Usual Care--Nurses telephoned patients 7 days prior to appointment to remind patients about scheduled GI appointment and to answer any questions.
- Total: Total of all reporting groups
Arm/Group | Usual Care | IVR3 | IVR7 | Total
Number analyzed (Participants) | 1199 | 1205 | 1206 | 3610
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.9) | 62.8 (10.2) | 62.5 (10.2) | 62.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 54 | 50 | 154
  Male | 1149 | 1151 | 1156 | 3456
Region of Enrollment [Number; unit: participants]
  United States | 1199 | 1205 | 1206 | 3610

OUTCOME MEASURES:

1. Primary Outcome: Appointment Nonadherence-colonoscopy
Description: Nonattendance was defined as canceling the colonoscopy appointment or not attending the appointment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | IVR3 | IVR7
Number analyzed (Participants) | 790 | 794 | 797
Participants | 348 | 333 | 303

2. Secondary Outcome: Nonattendance-flexible Sigmoidoscopy
Description: Nonattendance was defined as canceling the flexible sigmoidoscopy appointment or not attending the appointment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Interactive Voice Response 3 Days Prior: IVR3-Interactive voice response system was used to remind patients 3 days before a scheduled appointment and to educate them about preparation procedures for the appointment
- Interactive Voice Response 7 Days Prior: IVR7-Interactive voice response system was used to remind patients 7 days before a scheduled appointment and to educate them about preparation procedures for the appointment
Arm/Group | Usual Care With Nurse Phone Call | Interactive Voice Response 3 Days Prior | Interactive Voice Response 7 Days Prior
Number analyzed (Participants) | 409 | 411 | 409
Participants | 155 | 169 | 164

3. Secondary Outcome: Preparation Nonadherence-colonoscopy
Description: Preparation nonadherence assessed whether patients had adequately prepared their bowels to complete the colonoscopy procedure.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care With Nurse Phone Call: Usual Care--Nurses telephoned patients 7 days prior to appointment to remind patients about scheduled GI appointment and to answer any questions about bowel prep procedures.
- Interactive Voice Response 3 Days Prior: IVR3-Interactive voice response system was used to remind patients 3 days before a scheduled appointment and to educate them about bowel preparation procedures for the appointment
- Interactive Voice Response 7 Days Prior: IVR7-Interactive voice response system was used to remind patients 7 days before a scheduled appointment and to educate them about bowel preparation procedures for the appointment
Arm/Group | Usual Care With Nurse Phone Call | Interactive Voice Response 3 Days Prior | Interactive Voice Response 7 Days Prior
Number analyzed (Participants) | 790 | 794 | 797
Participants | 348 | 349 | 319

4. Secondary Outcome: Preparation Non-adherence-flexible Sigmoidoscopy
Description: Preparation nonadherence assessed whether patients had adequately prepared their bowels to complete the flexible sigmoidoscopy procedure.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care With Nurse Phone Call | Interactive Voice Response 3 Days Prior | Interactive Voice Response 7 Days Prior
Number analyzed (Participants) | 409 | 411 | 409
Participants | 164 | 173 | 168

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Groups:
- IVR7: Arm 2 (IVR3) included interactive voice response calls delivered to patients 7 days prior to the scheduled appointment. Calls were intended as appointment reminders and as interactive, but pre-recorded, opportunities for education on preparation procedures.
Arm/Group | Usual Care | IVR3 | IVR7
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes